CLINICAL TRIAL: NCT01110668
Title: Evaluation of Nilotinib In Patients With Advanced Gastrointestinal Stromal Tumor (GIST) Previously Treated With Imatinib
Brief Title: Evaluation of Nilotinib In Patients With Advanced Gastrointestinal Stromal Tumor (GIST)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CAMN107DTR01T
Record Dates: First submitted 2010-04-22; First posted 2010-04-27 (Estimated); Last update posted 2017-02-28 (Actual); Status verified 2017-02

CONDITIONS: Gastrointestinal Stromal Tumor
Keywords: Unresectable; metastatic gastrointestinal stromal tumor; disease progression; progression-free survival
MeSH Terms: conditions — Gastrointestinal Stromal Tumors; Disease Progression | interventions — nilotinib

ARMS (1):
- Nilotinib (Experimental)
  Interventions: Drug: Nilotinib

INTERVENTIONS:
Drug: Nilotinib

SUMMARY:
This study will assess time-to-disease progression in patients with advanced gastrointestinal stromal tumor (GIST) previously treated with imatinib ≥600 mg.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed diagnosis of GIST that is unresectable and/or metastatic
* Radiological confirmation of disease progression or intolerance to imatinib therapy at a any dose
* At least one measurable site of disease on CT scan at Visit-2
* WHO Performance Status of 0, 1 or 2 at Visit-2
* Patients must have normal organ, electrolyte, and marrow function at Visit-1 and Visit-2

Exclusion Criteria:

* Prior treatment with nilotinib or any other tyrosine kinase inhibitors except imatinib.
* Treatment with any cytotoxic and/or investigational cytotoxic drug ≤ 4 weeks
* Prior or concomitant malignancies other than GIST
* Impaired cardiac function at Visit-1 or 2
* Patients with severe and/or uncontrolled concurrent medical disease
* Use of therapeutic coumarin derivatives
* Use of any medications that prolong the QT interval
* Use of CYP3A4 inhibitors
* Patients who have undergone major surgery ≤ 2 weeks prior to Visit-1 or who have not recovered from side effects of such surgery
* Patients who have received wide field radiotherapy ≤ 4 weeks or limited field radiation for palliation < 2 weeks prior to Visit-1 or who have not recovered from side effects of such therapy

Other protocol-defined inclusion/exclusion criteria may apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2008-09; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
To evaluate time-to-disease progression in patients with advanced gastrointestinal stromal tumor (GIST) previously treated with imatinib ≥600 mg. | every 8 weeks

SECONDARY OUTCOMES:
To determine progression-free survival and the response rate of nilotinib in patients with advanced GIST previously treated with imatinib ≥600 mg. | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (4):
- Turkey (Türkiye) (4):
  - Novartis Investigative Site, Adana
  - Novartis Investigative Site, Ankara
  - Novartis Investigative Site, Istanbul
  - Novartis Investigative Site, Izmir